CLINICAL TRIAL: NCT01963871
Title: The Effect of Yoga in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yvonne Colgrove, PT, PhD (Other)
Responsible Party: Sponsor-Investigator, Yvonne Colgrove, PT, PhD, Clinical Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13763
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Low Back Pain
Keywords: chronic low back pain; low back pain; yoga
MeSH Terms: conditions — Low Back Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga in Chronic Low Back Pain (Experimental): 12 weeks of no yoga followed by 12 weeks of yoga, 2 times per week for individuals with chronic low back pain
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Twice weekly one hour sessions of Hatha Yoga for 12 weeks

SUMMARY:
The purpose of this study is to determine if yoga is an effective intervention in treating individuals with chronic low back pain (LBP).

DETAILED DESCRIPTION:
Chronic LBP is a major public health problem associated with functional and psychological disability. Conservative interventions are often prescribed to people suffering from chronic LBP, but alternative interventions like yoga are not well researched. The regulator practice of yoga may improve pain, disability or quality of life in people with chronic LBP.

Study participation will last approximately 24 weeks. Yoga sessions will last 12 weeks for 2 one hour sessions per week

ELIGIBILITY:
Inclusion Criteria:

* a history of chronic LBP with degenerative joint or disc disease > than 3 months (47-48)
* present with at least minimal pain (3 out on a 0 - 10 pain scale where 0 = no pain, 10 = maximum pain imaginable)
* disability (30% or more per Oswestry Disability Scale),
* score more than 24 on the Folstein Mini-Mental State Exam
* English comprehending individuals naïve to structured yoga practice

Exclusion Criteria:

* known current pregnancy
* claustrophobia
* glaucoma
* significant or chronic decline in immune function such as reported immune related diagnosis like pneumonia or systemic infection
* LBP resulting from something other than disc or joint disease
* spinal stenosis, spinal fusion or other orthopedic surgery in the past six months
* mental disease/psychosis such as dementia
* prior history of chronic neurological disorders (e.g. stroke, Parkinson's disease, multiple sclerosis)
* fibromyalgia
* radiculopathy
* standard MRI exclusion criteria
* inability to make regular time commitments
* no transportation means to the scheduled yoga sessions
* experience with regular practice of yoga within the past year.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
self-perceived pain and disability | Change in questionnaire scores from baseline to week 24
  perceived pain and disability as measured by the standard questionnaires of Numeric Rating Scale and Oswestry Disability Scale

SECONDARY OUTCOMES:
change in physical function | Change from baseline to week 24
  measured by changes in scores on standard tests of core strength, spinal range of motion and muscular flexibility
change in immunity | Change from baseline to week 24
  measured by serum immune markers

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States